CLINICAL TRIAL: NCT00032825
Title: A Phase I Trial of High Dose Ketoconazole Plus Weekly Docetaxel in Metastatic Androgen Independent Prostate Cancer
Brief Title: Ketoconazole Plus Docetaxel to Treat Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020149; 02-C-0149; NCT00039221 (obsolete NCT alias)
Record Dates: First submitted 2002-04-03; First posted 2002-04-04 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2012-05-04

CONDITIONS: Prostatic Neoplasms
Keywords: Combination; Microtubule; Hormonal; Chemotherapy; Pharmacokinetics; Prostate Cancer; Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: Ketaconazole
Drug: Docetaxel

SUMMARY:
This study will determine the maximum dose of docetaxel that can be given safely in combination with ketoconazole for treating advanced prostate cancer. Docetaxel is approved for the treatment of several other types of cancers; ketoconazole is an approved antifungal medication that is also commonly used in high doses to treat prostate cancer.

Patients 18 years of age and older with advanced prostate cancer that does not respond to hormone therapy may be eligible for this study. Candidates will be screened with blood tests to evaluate liver, kidney and other organ function and with x-rays, scans, or other imaging tests to determine the extent of disease.

Participants will take the following medications:

* Docetaxel daily, infused through a vein over 30 minutes, in 4-week cycles-3 consecutive weeks of drug followed by one week of rest
* Dexamethasone, 12 hours and 1 hour before and 12 hours after docetaxel infusions to help prevent fluid retention caused by the docetaxel
* Ketoconazole, 3 times a day
* Hydrocortisone, twice a day to replace a loss of natural steroids caused by the ketoconazole

Patients will be hospitalized 1 to 2 days each for the first and second doses of docetaxel to allow for frequent blood draws to measure blood levels of the drug. Ketoconazole will be started about 2 weeks after the first dose of docetaxel and the second dose of docetaxel will be given 2 days after that. In order to determine the maximum tolerated dose of docetaxel, the first few patients in the study will be given a low dose of the drug, and subsequent patients will get increasingly higher doses until unacceptable side effects occur. Because prostate cancer cells may grow if exposed to testosterone, patients may have to have their testosterone production suppressed either surgically (removal of the testicles) or medically with an injection of leuprolide or goserelin, which are luteinizing hormone-release hormone agonists that reduce the amount of testosterone.

Imaging studies, such as x-rays, bone scans or computed tomography (CT) scans, will be done about every 3 months to examine how the tumor is responding to therapy. After six treatment cycles, patients will have monthly chest x-rays to check for fluid around the lining of the lungs, which may occur as a result of docetaxel therapy.

Treatment is expected to continue for at least 3 to 6 months, although this time could be shortened or extended depending on the tumor response to therapy or side effects of the drugs. Patients who do not experience bad side effects and whose tumor does not grow during the first 3 treatment cycles will continue treatment; those who experience unacceptable side effects will be taken off the study.

...

DETAILED DESCRIPTION:
High dose ketoconazole and weekly docetaxel have both been shown to have activity against androgen independent prostate cancer (AIPC). We have demonstrated synergy in prostate cancer in an in vitro model. This is an open label phase I study of high-dose ketoconazole plus weekly docetaxel in patients with metastatic AIPC. The primary objective of this study will be to determine the side effect profile of ketoconazole when combined with weekly docetaxel therapy and determine the maximum tolerated dose (MTD) and a recommended phase II dose (RPIID) of docetaxel when combined with high dose ketoconazole. Since ketoconazole may alter the metabolism of docetaxel, this study will evaluate potential drug interactions and adverse events between these two agents. Ketoconazole dose will be 600mg per day (given 200 mg, three times a day), plus 30mg of hydrocortisone (20mg in the morning and 10mg in the evening), plus docetaxel 10-43 mg/m(2) in a dose escalation, repeated in 28-day cycles, comprising weekly treatments for three consecutive weeks followed by one week off. Each patient will be evaluated every four weeks for the duration of the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histopathological documentation of prostate cancer confirmed in the Pathology Department of the Clinical Center at the National Institutes of Health or the National Naval Medical Center prior to starting this study. Patients whose pathology specimens are no longer available may be enrolled in the trial, if the patient has a clinical course consistent with prostate cancer and pathologic documentation of the diagnosis.

Patients must have metastatic progressive androgen-independent prostate cancer (progressive prostate cancer while continuing to receive hormonal ablation, such as that of an LHRH agonist) documented prior to entry. Progression must be documented by at least one of the following parameters:

1. Two consecutively rising PSA levels, separated by at least one week, with at least one measurement that is 50% above the nadir reached after the last therapeutic maneuver (as long as the measurement is 5 ng/ml or greater); and/or,
2. At least one new metastatic deposit on Tc-99 bone scintigraphy; and/or,

Progression of soft tissue metastases as measured by appropriate modalities (i.e., imaging, palpation):

1. Development of new area of malignant disease (measurable or non-measurable);
2. Measurable disease progression by RECIST criteria;
3. At least 4 weeks off of flutamide and 6 weeks off of bicultamide and nilutamide.

Patients who have not undergone surgical castration must continue treatment with an LHRH agonist. If for some reason the LHRH agonist has been discontinued prior to entry on the study, then it should be reinstituted and disease progression must be documented.

Patients must have a life expectancy of more than 3 months.

Patients must have a performance status of 0 to 2 according to the ECOG criteria.

Patients must have recovered from any acute toxicity related to prior therapy, including surgery.

Hematological eligibility parameters (within 2 weeks before starting therapy):

1. Granulocyte count greater than or equal to 1,500/mm(3)
2. Platelet count greater than or equal to 100,000/mm(3)

Biochemical eligibility parameters (within 2 weeks before starting therapy):

1. If the creatinine is greater than 1.5 mg/dl, a 24 hour urine collection must be obtained, and measured creatinine clearance must be at least 40 mL/min.
2. Hepatic function: Hepatic: Bilirubin less than 1.0 mg/dl, AST and ALT less than 2.5 times upper limit of normal. If the alkaline phosphatase is greater than 2.5 times the upper limit of normal, it must be fractionated and the hepatic alkaline phosphatase should be less than 2.5 times the upper limit of normal.

Hormonal profile for patients with prostate cancer

1. All patients who have not undergone surgical castration must have a serum testosterone under 50 ng/ml and continue on their GnRh agonist.

Patients must not have other active malignancies (within the past two years with the exception of non-melanoma skin cancers or carcinoma in situ of the bladder).

Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), New York Heart Assoc. class II-IV congestive heart failure are not eligible.

Patients must be able to understand and sign an informed consent form.

Patients must be willing to travel from their home to the NIH for follow-up visits.

Patients must be greater than or equal to 18 years of age.

Must be able to ingest oral medications to be eligible.

EXCLUSION CRITERIA:

Patients with brain metastases will not be eligible.

Patients who have received strontium or samarium will not be eligible.

HIV-positive patients receiving combination anti-retroviral therapy will be excluded because of possible pharmacokinetic interactions with ketoconazole, docetaxel or other agents administered during the study. In fact, ketoconazole has been found to increase the toxic effects of several protease inhibitors by affecting CYP3A4 activity.

Patients on theophylline will be excluded.

Patients who are receiving cisapride will be excluded.

Patients who are receiving HMG-CoA inhibitors (lovastatin, atorvastatin, simvastatin, pravastatin and cerivastatin)

Patients currently taking known inhibitors and/or inducers of CYP3A4; patients taking known substrates of CYP3A4 will be evaluated by the primary investigator.

Patients who are receiving terfenadine, midazolam, triazolam, alprazolam, astemizole, loratadine, rifampin, isoniazid, dofetilide, pimozide, sirolimus or erythromycin will be excluded.

Because gastric acidity is necessary for the dissolution and absorption of ketoconazole, concomitant administration of drugs which decrease gastric acid output or increase gastric pH (e.g., antacids, cimetidine, ranitidine, antimuscarinics, omeprazole, and lansoprazole) may decrease absorption and thus will be prohibited.

Patients requiring warfarin will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2002-03-19; Study Completion 2011-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L Dahut, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bissery MC, Guenard D, Gueritte-Voegelein F, Lavelle F. Experimental antitumor activity of taxotere (RP 56976, NSC 628503), a taxol analogue. Cancer Res. 1991 Sep 15;51(18):4845-52. PMID 1680023
- [Background] Crawford ED, Eisenberger MA, McLeod DG, Spaulding JT, Benson R, Dorr FA, Blumenstein BA, Davis MA, Goodman PJ. A controlled trial of leuprolide with and without flutamide in prostatic carcinoma. N Engl J Med. 1989 Aug 17;321(7):419-24. doi: 10.1056/NEJM198908173210702. PMID 2503724
- [Background] Bubley GJ, Carducci M, Dahut W, Dawson N, Daliani D, Eisenberger M, Figg WD, Freidlin B, Halabi S, Hudes G, Hussain M, Kaplan R, Myers C, Oh W, Petrylak DP, Reed E, Roth B, Sartor O, Scher H, Simons J, Sinibaldi V, Small EJ, Smith MR, Trump DL, Wilding G, et al. Eligibility and response guidelines for phase II clinical trials in androgen-independent prostate cancer: recommendations from the Prostate-Specific Antigen Working Group. J Clin Oncol. 1999 Nov;17(11):3461-7. doi: 10.1200/JCO.1999.17.11.3461. PMID 10550143
- [Derived] Sissung TM, Danesi R, Kirkland CT, Baum CE, Ockers SB, Stein EV, Venzon D, Price DK, Figg WD. Estrogen receptor alpha and aromatase polymorphisms affect risk, prognosis, and therapeutic outcome in men with castration-resistant prostate cancer treated with docetaxel-based therapy. J Clin Endocrinol Metab. 2011 Feb;96(2):E368-72. doi: 10.1210/jc.2010-2070. Epub 2010 Nov 24. PMID 21106711